CLINICAL TRIAL: NCT01707498
Title: Clinical Evaluation of Brain-Computer Interface for Helping Communication of Quadriplegic Patients
Brief Title: Robust Intelligent Keyboard for Quadraplegic Patients
Acronym: PVCRoBIK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: University of Versailles (Other)
Responsible Party: Principal Investigator, david orlikowski, PROFESSOR, Centre d'Investigation Clinique et Technologique 805
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A00613-40
Record Dates: First submitted 2012-10-05; First posted 2012-10-16 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Quadraplegia
Keywords: BCI; TETRAPLEGIA; COMMUNICATION; P300; ASSISTIVE TECHNOLOGIE
MeSH Terms: conditions — Quadriplegia; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetraplegic patients (Experimental): Scanning device RoBIK Brain-Computer Interface
  Interventions: Procedure: Scanning device; Procedure: RoBIK Brain-Computer Interface
- Healthy volunteers (Experimental): RoBIK Brain-Computer Interface
  Interventions: Procedure: RoBIK Brain-Computer Interface

INTERVENTIONS:
Procedure: Scanning device — Patients will be asked to spell a text with a specific scanning device. The most appropriate contactor or clicking device will be chosen by a senior therapist.
  Arms: Tetraplegic patients
Procedure: RoBIK Brain-Computer Interface — Patients will be asked to spell a text with the BCI

SUMMARY:
This is multi-center prospective randomized trial evaluating the effectiveness of a new brain-computer interface for communication of quadriplegic patients in a clinical context. This performance of this will compared to traditional assistive technology (scanning system) and to performance of a healthy volunteer population.

DETAILED DESCRIPTION:
The evaluation aims to estimate the performance of BCIs in patient and healthy subjects in a clinical setting (primary objective) and to compare this performance with an existing assitive technology adapted to the target population of this study (scanning system). A quadriplegic patient population (n = 10) evaluated the two techniques and a population of healthy subjects (n = 10) evaluated the BCI only.

When a subject meets all the eligibility criteria and is not discarded by any non-inclusion criteria, he is included in the study. The order of the two techniques to be compared is randomized.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Informed consent
* Adults aged more than 18yo
* Passed complete medical check-up (heart-rate, blood pressure,...)
* Negative pregnancy test

Quadripleagic patients:

* Informed consent
* Adults aged more than 18years
* Passed medical exam
* Negative pregnancy test
* Full medical checkup
* haemodynamic stability

Exclusion Criteria:

Healthy volunteers:

* history of epilepsy or seizure
* auditory or visual deficit
* atopic scalp dermatitis
* hypersensitivity to gold
* curator/guardianship/under protection of judicial authority
* unable to understand the information note and/or to cooperate
* no social security
* can't read

Quadripleagic patients:

* history of epilepsy or seizure
* auditory or visual deficit
* cerebral lesion
* atopic scalp dermatitis
* hypersensitivity to gold
* curator/guardianship/under protection of judicial authority
* unable to understand the information note and/or to cooperate
* no social security
* can't read
* included in a different clinical trial with exclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
BIT RATE IN BIT PER MINUTE(bpm) | 15 MINUTES
  Bitrate (bpm): transfer of information from patient to computer in bits per minutes. This is a reference measurement to compare P300 speller Brain Computer Interfaces. It uses: number of choices on the interface (N), the average time to select one key (t) and the error rate (e)

SECONDARY OUTCOMES:
Installation time (seconds) | 60 mns
  Installation time (seconds), Number of caracters spelt in a pre-defined time, Error rate: Area Under the Receiver Operating Curve (AUROC), Balanced Error Rate (BER), Visual Analogous Scale for tiredness (before, after the use) and overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: LOUIS MAYAUD, ENGINEER, Study Director — CIC IT 805
Locations (1):
- Hopital Raymond Poincare, Garches, France